CLINICAL TRIAL: NCT00842985
Title: Dronabinol Interactions in Humans
Brief Title: Dronabinol Interactions With Cognitive Enhancing Drug in Humans
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: VA Office of Research and Development (U.S. Federal Agency); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Mehmet Sofuoglu, M.D., Ph.D., Yale University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 0702002357; MIRECC 00000000 (Registry Identifier: Veteran's Administration); P50DA009241 (NIH)
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Results first posted 2012-12-17 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-04

CONDITIONS: Cannabis; Marijuana Abuse
Keywords: Cannabis Abuse; Cannabis Dependence; Cannabis-Related Disorder; Marijuana Dependence; Marihuana Abuse
MeSH Terms: conditions — Marijuana Abuse | interventions — Dronabinol; Modafinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- drug condition (Other): Participants received each drug condition in sequential order across 4 test days. Not all participants received the interventions in the same order.
  Interventions: Drug: drug condition

INTERVENTIONS:
Drug: drug condition — Dronabinol (15mg) or Modafinil (400mg) or Dronabinol + Modafanil or placebo
  Other Names: Marinol, Provigil,

SUMMARY:
Marijuana use is a major problem among veterans and non-veterans. A patient's use of marijuana while engaged in psychotherapy treatment may affect their memory and, therefore, limit their ability to benefit from treatment. This study is designed to test a new pharmacotherapy, modafinil, which has the potential to improve memory functioning in marijuana using individuals.

We hypothesize that modafinil treatment will decrease ratings of drug liking and improve cognitive measures, especially episodic memory.

DETAILED DESCRIPTION:
The impairment of episodic memory in marijuana abusers has important treatment implications. Since many treatments, including cognitive-behavioral therapy, strongly utilize episodic memory, marijuana use during treatment may lead to diminished treatment outcomes. In addition, lessened response inhibition may lead to elevated rates of drug relapse while in treatment. Consequently, a treatment which will improve episodic memory and response inhibition may lead to improved treatment outcomes in marijuana users. One such treatment is modafinil.This study will be a 4 session within-subjects, double-blind, crossover study evaluating the impact of modafinil (400 mg/day) on the cognitive, subjective, and physiological effects of marijuana. Across 4 sessions, subjects will be randomly assigned to receive either oral placebo, modafinil (400mg), dronabinol (15mg), or dronabinol and modafinil. Outcome measures will include physiological, cognitive, and subjective drug effects.

Currently this study complete and has been published.

ELIGIBILITY:
Inclusion Criteria:

* • Males and females between 18 and 55 years old will be eligible for this study.

  * Marijuana used at least once in last 2 months and at least 10 times in lifetime.
  * Subjects do not meet DSM-IV criteria for marijuana abuse or dependence.
  * Subjects are NOT seeking treatment for substance abuse or dependence.
  * Females must not be pregnant as determined by pregnancy screening, nor breast feeding, and must be using acceptable birth control methods other than oral contraceptive pills (OCP). Modafinil may cause OCP to be ineffective. Acceptable forms of birth control are condoms, diaphragms, and IUDs.
  * No alcohol or drugs 24 hours prior to testing session.
  * Subjects must agree to not drive to or from session.

Exclusion Criteria:

* • History of heart disease, left ventricular hypertrophy, ischemic ECG changes, chest pain, arrhythmia, hypertension.

  * History of severe renal or hepatic diseases.
  * History of psychosis, schizophrenia or bipolar type I disorder.
  * History of seizure disorder.
  * Current diagnosis of alcohol and other drug dependence (other than nicotine).
  * A positive urine toxicology result for cocaine or opiates at intake.
  * Current use of over-the-counter or prescription psychoactive drugs (antidepressant, anxiolytics, antipsychotics, mood stabilizers, psychostimulants).
  * Liver function tests (ALT or AST) greater than 3 times normal.
  * Known allergy to modafinil or dronabinol.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2008-09; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sofuoglu, M.D,Ph.D., Principal Investigator — Yale University
Locations (1):
- Department of Veterans Affairs Hospital, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sugarman DE, Poling J, Sofuoglu M. The safety of modafinil in combination with oral ∆9-tetrahydrocannabinol in humans. Pharmacol Biochem Behav. 2011 Mar;98(1):94-100. doi: 10.1016/j.pbb.2010.12.013. Epub 2010 Dec 21. PMID 21176784
- [Derived] Bosnjak Kuharic D, Markovic D, Brkovic T, Jeric Kegalj M, Rubic Z, Vuica Vukasovic A, Jeroncic A, Puljak L. Cannabinoids for the treatment of dementia. Cochrane Database Syst Rev. 2021 Sep 17;9(9):CD012820. doi: 10.1002/14651858.CD012820.pub2. PMID 34532852

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: There were 4 sessions given in a counterbalanced order: Dronabinol+Modafinil, Dronabinol+Placebo, Placebo+Modafinil, Placebo+Placebo.
  Not all participants received the interventions in the same order.
Period: Screening
Arm/Group | All Participants
Started | 53
Completed | 26
Not Completed | 27
Not completed — Did not meet entrance requirements | 27
Period: First Intervention
Arm/Group | All Participants
Started | 26 (Signed Consent)
Completed | 20 (Completed 1st Intervention)
Not Completed | 6
Not completed — Withdrawal by Subject | 3
Not completed — Protocol Violation | 3
Period: Washout Period of GE 4 Days
Arm/Group | All Participants
Started | 20
Completed | 18
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Second Intervention
Arm/Group | All Participants
Started | 18
Completed | 17
Not Completed | 1
Period: Washout Period of GE 4 Days
Arm/Group | All Participants
Started | 17
Completed | 15
Not Completed | 2
Not completed — Withdrawal by Subject | 2
Period: Third Intervention
Arm/Group | All Participants
Started | 15
Completed | 15
Not Completed | 0
Period: Washout Period of GE 4 Days
Arm/Group | All Participants
Started | 15
Completed | 15
Not Completed | 0
Period: Fourth Intervention
Arm/Group | All Participants
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 53
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.7 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 53

OUTCOME MEASURES:

1. Primary Outcome: CANTAB:CAmbridge Neuropsychological Test Automated Battery RVIP: Rapid Visual Information Processing
Description: CANTAB RVIP is one component of this computerized battery and is a measure of sustained attention with a working memory component.
  This study used two subscales of the RVIP.
  1. RVP A' ( Target sensitivity, a measure of the ability to detect sequences.) The range is from 0-1; bad to good.
  2. RVP B'' ( Response bias, which is a measure of the tendency to respond regardless of whether a target is present.
  The range is from -1 to +1 ; bad to good
  The numbers represent probabilities as units on a scale.
Time Frame: Once for each test session (4 total).
Population: Subjects who completed all four treatment sessions. Three of these 15 subjects were not analyzed due to validity concerns of the cognitive data for at least one of the four testing sessions.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- THC+Modafinil: Session where THC+Modafinil was given.
- THC+Placebo: Session where TCH and Placebo Modafinil were given
- Pla+Modafinil: Session where Placebo THC and Modafinil were given
- Placebo+Placebo: Session where placebo THC and Placebo Modafinil were given.
Arm/Group | THC+Modafinil | THC+Placebo | Pla+Modafinil | Placebo+Placebo
Number analyzed (Participants) | 12 | 12 | 12 | 12
units on a scale | 0.91 (.1) | 0.9 (.1) | 0.92 (.1) | 0.9 (.1)

ADVERSE EVENTS:
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 0/26
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
One dose of modafinil Brief treatment duration and use of a low dose of THC Cognitive testing assessed only two tasks. Outcome measures were limited by small sample size.

Limited generalizability because heavy cannibas users were excluded

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No